CLINICAL TRIAL: NCT04448990
Title: Antinociceptive Effect of Transauricular Electrical Vagal Nerve Stimulation and Its Underlying Mechanisms
Brief Title: Antinociceptive Effect of Transauricular Electrical Vagal Nerve Stimulation
Acronym: TVNS_TSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BB 196/18
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Two periods (real and sham tVNS) randomized crossover investigation in healthy volunteers
Who Masked: Participant, Outcomes Assessor
Masking Description: Real tVNS will be applied using pre-defined characteristics of tVNS device to cymba conchae of the auricle, sham procedure will be the same, however applied to tubule of the auricle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tVNS (Experimental): Stimulation will be applied using TENS device eco 2 (Schwa-Medico, Pierenkemper GmbH, Ehringshausen, Germany) bilaterally at the cymba conchae of the auricles for 20 minutes. Current intensity (1-max. 10 mA) will be individually adjusted for each ear separately until the maximal tVNS intensity, which is not uncomfortable or painful, will be achieved.
  Interventions: Device: TENS eco 2 Transauricular vagal nerve stimulation
- Sham (Sham Comparator): Same stimulation will be applied using TENS device eco 2 (Schwa-Medico, Pierenkemper GmbH, Ehringshausen, Germany) to bilaterally to the earlobes for 20 minutes. Current intensity (1-max. 10 mA) will be individually adjusted for each ear separately until the maximal tVNS intensity, which is not uncomfortable or painful, will be achieved.
  Interventions: Device: Sham TENS eco 2

INTERVENTIONS:
Device: TENS eco 2 Transauricular vagal nerve stimulation — Auricular electrical stimulation will be applied bilaterally using Transcutaneous Electrical Nerve Stimulation device TENS eco 2 (Schwa-Medico, Pierenkemper GmbH, Ehringshausen, Germany).
  tVNS will be applied bilaterally using electrical square impulses delivered in blocks of 9 impulses with a frequency of 100 Hz and a pulse width of 200 μs emitted twice per second resulting in mixed frequency pattern of 100 Hz/2 Hz with the current intensity, that will be individually adjusted for each ear separately until the maximal tVNS intensity, which is not uncomfortable or painful, will be achieved.
  Arms: tVNS
Device: Sham TENS eco 2 — Sham
  Arms: Sham

SUMMARY:
This investigation is going to study whether electrical tVNS applied at the cymba of auricular conchae reduces central sensitization of experimentally induced pain in comparison with electrical sham stimulation applied at the earlobes and whether the hypoalgesic effects of tVNS disappear after pharmacological block of muscarinic receptors. Also, this investigation will examine whether tVNS is associated with activation in brain areas, involved in processing of thermal pain stimuli and emotional and vegetative modulation of thermal pain in subjects who will respond with antinociceptive reaction to tVNS.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged 18-45 years old, who have given informed consent
* at least two days free from consume of recreational drugs
* no local infection at the site of tVNS and pain stimulation

Exclusion Criteria:

* psychiatric disorders
* abnormal skin conditions (infection, scars, psoriasis, eczema) at the site of tVNS
* contra-indications for MRI (e.g. claustrophobia, pregnancy, tattoos, metallic implants)
* history of coronary heart disease, cardiac arrhythmia, glaucoma, allergy to sulphates

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Unpleasantness of pain | Continuously 5 minutes during the experimental heat pain stimulation
  perceived unpleasantness of pain, which participants will rate continuously during the repetitive heat stimulation using a computerized visual analogue scale (CoVAS, Medoc Advanced Medical Systems, Ramat Yishai, Israel) ranging from 0 (= not unpleasant at all) to 100 (= intolerable pain).

SECONDARY OUTCOMES:
Heart rate | Continuously 5 minutes during the experimental heat pain stimulation
  Heart rate (bpm)
Blood pressure | 4 times during 5 minutes of the experimental heat pain stimulation
  Systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available of request